CLINICAL TRIAL: NCT00822679
Title: Eszopiclone and Inflammatory Mediators in Patients With Acute Coronary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry); Southern Arizona VA Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sairam Parthasarathy, Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HSC# 07-0797-01
Record Dates: First submitted 2009-01-12; First posted 2009-01-14 (Estimated); Results first posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-10

CONDITIONS: Acute Coronary Syndrome; Sleep Disorder
Keywords: Acute Coronary Syndrome; cytokines; pro-coagulant mediators; sleep disorders
MeSH Terms: conditions — Acute Coronary Syndrome; Sleep Wake Disorders | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Eszopiclone (Experimental): Subjects receive Eszopiclone for three consecutive nights to observe changes in sleep measures, and inflammatory and coagulation factors
  Interventions: Drug: Eszopiclone
- 2: Placebo (Placebo Comparator): Subjects given placebo for 3 consecutive nights to observe changes in sleep measures, and inflammatory and coagulation factors
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Eszopiclone — Subject receives Eszopiclone for 3 consecutive nights. 3 mg orally at bedtime for patients age 64 and under, and 2 mg QHS for patients age 65 and older.
  Other Names: Lunesta
  Arms: 1: Eszopiclone
Other: Placebo — Subjects are given placebo for 3 consecutive nights
  Arms: 2: Placebo

SUMMARY:
The purpose of the study is to examine the effects of Eszopiclone, a sleep aid, on inflammatory mediators and coagulability in patients with a recent myocardial infarction.

DETAILED DESCRIPTION:
Abnormalities of sleep are common in hospitalized patients, but the mechanisms and consequences are not well understood. In many of these patients, sleep is very disrupted, occurs during the daytime, and circadian rhythm is diminished or lost. Hospitalized patients experience more frequent arousals and awakenings than is normal and show decreases in rapid eye movement and slow wave sleep. The degree of sleep fragmentation is at least equivalent to that seen in patients with obstructive sleep apnea. About 20% of arousals and awakenings are related to noise, 10% are related to health care personnel and care-related activities, and the cause for the remainder is not known, although severity of underlying disease is likely an important factor.

In studies of sleep following acute myocardial infarction, marked disturbances have been found in patients, whether in the ICU and on the wards. These disturbances include long periods of wakefulness; poor sleep efficiency, and disruption of REM sleep. The fact that there is also a loss in circadian rhythm in these patients may indicate a widespread disruption of bodily homeostasis which, in turn, may be related to the infarct itself, to a more generalized physiological response to stress or to other factors. Sleep disruption can induce sympathetic activation and elevation of blood pressure, which may contribute to patient morbidity.

It has been shown that there is an increased level of some inflammatory and coagulation factors in the recovery period following an acute myocardial infarction (MI). Post MI patients have higher levels of TNF-α, IL-6 and tissue plasminogen activator as well as lower levels of antithrombin III and protein C.

The aim of this study is to determine whether the sleep-aid Eszopiclone can improve sleep, decrease inflammation, and decrease pro-coagulation factors in patients who have recently suffered myocardial infarction when compared with a control group without sleep aids. Eszopiclone is a benzodiazepine receptor agonist which improves sleep quality by reducing the time to sleep onset and reduces wakefulness during the sleep period. Unlike benzodiazepines, it does not affect the deeper stage 3 and 4 sleep. The result is that it provides a more nearly normal night sleep than other sleep aids. It is hoped that improved sleep patterns will result in more rapid normalization of inflammatory and coagulation factors and perhaps more rapid recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recent (less than or equal to 8 weeks) "uncomplicated" acute myocardial infarction, can either be ST elevation MI (STEMI) or non-ST elevation MI (non-STEMI) and subsequent to successful treatment (percutaneous revascularization or medical therapy).

Exclusion Criteria:

* Obstructive sleep apnea (OSA, defined as apnea-hypopnea index > 15 per hour) or previous diagnosis of OSA.
* Patients with life-threatening arrhythmias (such as atrial fibrillation/flutter with hypotension, ventricular tachycardia, or ventricular fibrillation, or significant heart block that requires pacing [Type III, Type IIb]), cardiogenic shock, severe heart failure requiring high levels of inspired oxygen (FiO2 >40%), persistent chest pain despite medical or other interventions, and patients who are considered too unstable to participate for other medical reasons or complications (such as concomitant strokes, retroperitoneal hematoma, gastro-intestinal bleeding). Also excluded are patients with history of cardiac arrest during the same hospitalization.
* Unable to take oral medications
* Use of other sedative-hypnotics
* Hypersensitivity to Eszopiclone or any component of the formulation
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sairam Parthasarathy, MD, Principal Investigator — Southern Arizona VA Health Care System
Locations (1):
- Southern Arizona VA Health Care System, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants screen failed. There was no subject randomized (n=0).
Period: Overall Study
Arm/Group | 1: Eszopiclone | 2: Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Eszopiclone | 2: Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Gender
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Changes in Circulating Inflammatory Cytokines (Interleukin [IL]-1B, IL-6, IL-10, and Tumor Necrosis Alpha [TNF-α]) and Pro-coagulant Mediators (Soluble P-selectin and CD40 Ligand).
Description: Not performed. Zero subjects were randomized. Many potential participants screen-failed.
Time Frame: 2 days
Population: Not performed. Zero subjects were randomized. Many potential participants screen-failed.
Arm/Group | 1: Eszopiclone | 2: Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Changes in Objective and Subjective Measures of Sleep
Time Frame: 4 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | 1: Eszopiclone | 2: Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Zero subjects were randomized. Many potential participants screen-failed. Study was closed due to difficulty with recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No